CLINICAL TRIAL: NCT00977262
Title: Effects of Fatty Acids on Postprandial Inflammatory Response of Healthy Obese and Type 2 Diabetic Obese Subjects
Brief Title: Postprandial Inflammation and Fatty Acids
Acronym: PIFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Dutch Diabetes Research Foundation (Other)
Responsible Party: Wageningen University, Division of Human Nutrition, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: NL2800108109
Record Dates: First submitted 2009-09-11; First posted 2009-09-15 (Estimated); Last update posted 2010-04-21 (Estimated); Status verified 2010-04

CONDITIONS: Cardiovascular Disease; Diabetes Type 2; Obesity
Keywords: fatty acids; peripheral blood mononuclear cells; inflammation; nutrigenomics
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Obesity; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Healthy control subjects, High saturated fat shake (Experimental)
  Interventions: Other: High saturated fat shake
- Healthy control subjects, High Monounsaturated fat shake (Experimental)
  Interventions: Other: High monounsaturated fat shake
- Healthy control subjects, High Polyunsaturated fat shake (Experimental)
  Interventions: Other: High polyunsaturated fat shake
- Healthy obese subjecs, High saturated fat shake (Experimental)
  Interventions: Other: High saturated fat shake
- Healthy obese subjects, High monounsaturated fat shake (Experimental)
  Interventions: Other: High monounsaturated fat shake
- Healthy obese subjects, High polyunsaturated fat shake (Experimental)
  Interventions: Other: High polyunsaturated fat shake
- Obese diabetes type 2 subjects, High Saturated fat shake (Experimental)
  Interventions: Other: High saturated fat shake
- Obese diabetes type 2 subjects, High Monounsaturated fat shake (Experimental)
  Interventions: Other: High monounsaturated fat shake
- Obese diabetes type 2 subjects, High polyunsaturated fat shake (Experimental)
  Interventions: Other: High polyunsaturated fat shake

INTERVENTIONS:
Other: High saturated fat shake — milkshake containing 95 gram of fat, high percentage of saturated fat
  Arms: Healthy control subjects, High saturated fat shake; Healthy obese subjecs, High saturated fat shake; Obese diabetes type 2 subjects, High Saturated fat shake
Other: High monounsaturated fat shake — milkshake containing 95 gram of fat, high percentage of monounsaturated fat
  Arms: Healthy control subjects, High Monounsaturated fat shake; Healthy obese subjects, High monounsaturated fat shake; Obese diabetes type 2 subjects, High Monounsaturated fat shake
Other: High polyunsaturated fat shake — milkshake containing 95 gram of fat, high percentage polyunsaturated fat
  Arms: Healthy control subjects, High Polyunsaturated fat shake; Healthy obese subjects, High polyunsaturated fat shake; Obese diabetes type 2 subjects, High polyunsaturated fat shake

SUMMARY:
The main objective is to elucidate the acute effects of an oral intake of either saturated, monounsaturated or polyunsaturated fatty acids on peripheral blood mononuclear cells (PBMC) whole genome expression of obese and type 2 diabetic obese subjects.

DETAILED DESCRIPTION:
Consumption of high-fat diets can lead to postprandial dyslipidemia, impairment of endothelial function, activation of immune cells and changes in gene expression profiles of immune cells such as peripheral blood mononuclear cells (PBMC). Recently it was shown that postprandial gene expression profiles of PBMC and plasma triglyceride (TG) and free fatty acid (FFA) responses are dependent on the type of dietary fat consumed (i.e. saturated, monounsaturated and polyunsaturated). Since obese and diabetic subjects usually are in a pro-inflammatory state and have dyslipidemia and endothelial dysfunction we are interested in the effect of different fatty acids in a high load on the PBMC gene expression profiles, plasma cytokine profiles and endothelial function of these subjects.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* male gender
* 50-70 yrs

For diabetic patients only:

* BMI >30 kg/m2
* Well-controlled diabetes: fasting plasma glucose concentration must be <10.0 mmol/l at the time of screening.
* Must be on sulphonylurea- or metformin therapy for at least 6 months with a constant dose for at least two months, or on dietary treatment for at least 6 months2.

For obese controls only:

* BMI > 30 kg/m2
* normoglycemic according to WHO criteria (OGTT, fasting blood glucose< 7 mmol/L, after 2 hr <7.8mmol/L)

For lean controls only:

* BMI 18-25 kg/m2
* normoglycemic according to WHO criteria (OGTT, fasting blood glucose< 7 mmol/L, after 2 hr <7.8mmol/L)

Exclusion Criteria:

For all participants:

* Female gender
* Age below 50 or above 70 years
* Hemoglobin levels <8.4 mmol/L
* Allergic to cow milk or dairy products
* Allergic to fish oil
* Vegetarian
* Tobacco smoker
* Current or recent (<4 weeks) use of fish oil supplements or more then four times fish/week; 24.35 g of EPA-DHA of fish per month (800 mg/day) as judged by the questionnaire.
* Received inoculations within 2 months of starting the study or planned to during the study
* Donated or intended to donate blood from 2 months before the study till two months after the study
* Unstable body weight (weight gain or loss > 3 kg in the past three months)
* Medical condition that can interfere with the study outcome (i.e. cardiovascular disease, gastrointestinal disease, renal dysfunction)
* Use of medications know to interfere with glucose homeostasis (i.e. corticosteroids)
* abuse of drugs and/or alcohol
* participation in another biomedical study within 1 month before the first screening visit

For obese, type 2 diabetic subjects only:

* severe diabetes which requires application of insulin
* diabetes-related complications

For obese subjects and lean controls only:

* hyperglycemic according to WHO criteria (OGTT, fasting blood glucose >6.0mM, after 2 hr>11mM)
* systolic blood pressure >160 mmHg or diastolic blood pressure > 100 mmHg
* Urinary glucose concentrations (>0.25 g/l)

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
PBMC gene expression profiles | 0, 2, 4 hrs

SECONDARY OUTCOMES:
PBMC inflammatory response capacity | 0, 2, 4 hrs
Endothelial function | 0, 2, 4 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Michael Muller, Prof, Study Chair — Chair Department of Human Nutrition NMG group; Lydia A Afman, PhD, Principal Investigator — Senior scientist department Human Nutrition Wageningen University
Locations (2):
- Netherlands (2):
  - Wageningen University, Division of Human Nutrition, Wageningen, Gelderland
  - Wageningen University, Division of Human Nutrition, Wageningen

REFERENCES:
- [Derived] Esser D, van Dijk SJ, Oosterink E, Muller M, Afman LA. A high-fat SFA, MUFA, or n3 PUFA challenge affects the vascular response and initiates an activated state of cellular adherence in lean and obese middle-aged men. J Nutr. 2013 Jun;143(6):843-51. doi: 10.3945/jn.113.174540. Epub 2013 Apr 24. PMID 23616512
- [Derived] van Dijk SJ, Mensink M, Esser D, Feskens EJ, Muller M, Afman LA. Responses to high-fat challenges varying in fat type in subjects with different metabolic risk phenotypes: a randomized trial. PLoS One. 2012;7(7):e41388. doi: 10.1371/journal.pone.0041388. Epub 2012 Jul 23. PMID 22844471